CLINICAL TRIAL: NCT05921942
Title: The Impact of Metformin Administration on the Clinical Outcome of Stage IV Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Sayed Abdelhafeez, Teaching Assistant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 262
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: metformin; Colorectal cancer; FOLFOX
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Patients who fulfill the inclusion criteria will be recruited and randomized into one of two groups:
  Group A: Patients will receive standard therapy FOLFOX PROTOCOL Group B: Patients will receive metformin (500 mg twice daily or 1000 mg once daily) on top of standard therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (No Intervention): Patients will receive standard therapy FOLFOX/XELOX PROTOCOL
- Group B (Active Comparator): Patients will receive metformin (500 mg twice daily or 1000 mg once daily) in addition to standard therapy FOLFOX/XELOX PROTOCOL
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500 mg twice daily or 1000 mg once daily
  Arms: Group B

SUMMARY:
Design: Prospective, randomized controlled trial Setting: Clinical Oncology and Nuclear Medicine, Ain Shams University Condition: Colorectal cancer

Patients will be randomized into one of two groups:

Group A: Patients will receive standard therapy FOLFOX PROTOCOL Group B: Patients will receive metformin (500 mg twice daily or 1000 mg once daily) on top of standard therapy

Assessment:

Baseline Assessment:

* Patient Full History: Age, sex, smoking history, occupational history, medical history, concurrent diseases and medications.
* Laboratory data:
* Complete blood test
* Liver functional test
* Renal function test
* Inflammatory Markers: Interleukin (IL)-6

EVERY 3 MONTH: CT/MRI /PET scan to detect the response to chemotherapy and progression , Quality of life by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30. (EORTC QLQC30), Assessment of chemotherapy toxicity using CTACE 4.0 .

Every 2 CYCLE: Lab examination (CBC, Liver function, Kidney function),CTACE SIDE EFFECTS EXAMINATION AFTER 6 MONTH : iL-6 LEVELS AFTER 1 YEAR : PFS AND OS

DETAILED DESCRIPTION:
Colon cancer is significant Public health problem and one of the most common cancers worldwide. With Annually, more than 1.36 million patients are diagnosed with this disease. Approximately, 694,000 colon cancer - associated mortalities Occur per year accounting for 8.5% of all cancer-related deaths and making colorectal cancer (CRC) the third most common cause of death.

Multiple risk factors for colon cancer were identified including increasing age, smoking, black race, obesity, low fiber and rich processed food diet or as so called western diet, insulin resistance, obesity, type 2 diabetes and the metabolic syndrome. (Kaneko et al.,2014).

Increased body weight and type 2 diabetes have been linked to many types of cancer. This association has primarily been attributed to insulin resistance and cluster factors of metabolic syndrome thought to also play additive carcinogenic roles. (Inoue and Tsugane, 2012). Diabetes, in specific, has been proposed as a risk factor for many cancers, including colon, breast, prostate, kidney, and pancreatic cancers (Giovannucii et al, 2010), (SteinmausC et al, 2011). Insulin resistance in patients with diabetes can pro-mote tumorigenesis by increasing the levels of insulin-like growth factor 1, steroidal sex hormones, and inflammation (Jaiving M, 2010). In addition, the So-Called-Western diet, rich in processed foods and meats, sedentary lifestyle and obesity are may be mediated by hyperinsulinemia. (Inoue and Tsugane, 2012).

Glucose, The Co- factor in all risk factors, is one source of energy for tumor cells to support its growth and proliferation. Tumor cells depend on the intake of amino acids such as glutamine. Glucose uptake is regulated by growth factor signaling in normal on-proliferating cells. Activation of growth factor receptors stimulates changes in intracellular signaling, which in turn modifies metabolic pathways in support of proliferative growth. Hyperglycemia is often wrongly implicated as the sole source of cancer nutrition in patients with diabetes, when in fact cancer cells can thrive using other energy sources promoted by genetic mutations and aberrant intracellular signaling (Handelsman et al., 2013). Insulin has been shown to affect the growth of both normal and neoplastic epithelial cells and to have the capability of promoting mitosis in vitro, directly or indirectly via Insulin-like growth factor 1 (IGF-1). It has been proposed that insulin and insulin-like growth factors may be involved in colon carcinogenesis (Trevisan et al., 2001), Aleksandrova et al., 2011). Insulin acts as a growth factor, and insulin receptors are present in normal and malignant colorectal cells. This action would be potentiated by hyperglycemia which induces the secretion of insulin (Trevisan et al., 2001). That was proven through Several studies have shown that abnormal glucose metabolism is associated with an increased risk of colon cancer (Khaw et al., 2004; Hsu et al., 2012).

The primary treatment of colon cancer in several stages is to surgically remove part of the colon or all of it (colectomy). however, most cases need chemotherapy after surgery to improve the likelihood of being cured especially if colon cancer has spread to nearby lymph nodes. Radiation therapy is also available after surgery, but it mainly does not improve cure rates in people with colon cancer, And more frequently for people with rectal cancer. In patients with stage III colon cancer, the addition of oxaliplatin to a regimen of 5-FU and LV is known as FOLFOX, which has become the adjuvant gold standard therapy. As for patients have not received any previous chemotherapy for metastatic disease, several studies were made where the expert opinion is that chemotherapy FOLFOX or CAPOX is recommended. (Goldberg, R. M. (2006) Metformin is known as a hypoglycemic agent that regulates glucose homeostasis by inhibiting liver glucose production and increasing muscle glucose uptake. In addition, it's the first line oral therapy used in the treatment of type II diabetes. During the past decade, there has been an increasing interest in the relationship between metformin and Colon cancer, including Onset and prognosis. In some studies, metformin may have anticancer effects both in vivo and in vitro settings Various mechanisms have been proposed for the anticancer effects of metformin. Several basic studies have demonstrated that metformin inhibits cancer cell proliferation, metabolism and angiogenesis by activating adenosine monophosphate-activated protein kinase (AMPK). AMPK plays a critical role in maintaining cellular functions under energy-restricted conditions. Activated AMPK inhibits the synthesis of glucose, lipids, proteins, and cell growth under general conditions (Dowling RJ, 2007), (Zakikihani M ,2006). It also, inhibits mTOR (mammalian target of rapamycin) signaling, subsequently inhibiting protein synthesis and cell proliferation, which may be a direct mechanism driving metformin-mediated suppression of cancer cell growth. Several other anticancer mechanisms have been proposed, including inhibition of serum insulin and insulin like growth factor 1 levels (Kalaany NY,2009) that In states of insulin resistance, works in the liver by lowering systemic glucose levels and improving secondary hyperinsulinemia, preventing the latter's effects on tumor growth and progression (Pollak MN , 2012 ) , downregulation of cyclin D1 protein expression(Bensahra I,2008), activation of apoptotic pathways (Isakovic A , 2007) , reversing the effects of the high-energy diet in promoting the growth of colon cancer by inhibiting expression of fatty acid synthase (Algirec , 2010) Although several mechanisms have been identified, it is necessary to determine other unknown antitumor mechanisms of metformin to identify appropriate cancer targets. A recent study, found that metformin treatment reduced interleukin 6 (IL-6) inflammatory, and epithelial mesenchymal transition (EMT) signaling using high-throughputdata, and then test the mechanism experimentally through human cell lines invitro (Kang et al, 2018). However, a study about metformin effect on IL-6 pathway clinically have never been addressed.

With Colon cancer, several clinical and preclinical studies about metformin preventive and antitumor effect have been performed. However, most studies are small and retrospective, and have evaluated the antitumor effects of metformin specifically in cancer patients with concurrent diabetes. Some of these studies have shown that diabetic patients with colon cancer who receive therapy with metformin had improved outcomes. A retrospective Korean study of 595 diabetic patients with stage I to IV CRC demonstrated that those who received metformin had a 3-year overall survival (OS) rate of 89.6 versus87.9% (P 1⁄4 .018) and 3-year CRC-specific survival rates of 92.4%versus 90.8% (P 1⁄4 .042) compared to those who did not receivemetformin.2 After adjusting for age, sex, body mass index (BMI), insulin therapy, use of other sulfonylureas, disease stage, aspirin use, and duration of diabetes, receipt of metformin and early tumor stage remained independent favorable prognostic factors for CRC-specific mortality. Another retrospective study of diabetic patients with CRC of all stages found a median OS of 76.9 months among metformin recipients versus 56.9 months among those who did not receive metformin (P 1⁄4 .048); again, after adjusting for possible confounding factors, type 2 diabetic patients treated with metformin were found to have a 30% relative improvement in OS compared to diabetic patients treated with other antidiabetic agents. A meta-analysis and a population-based study showed that the use of metformin among diabetic patients decreased the risk of developing CRC. The meta-analysis of published data from retrospective and case control studies, which included 108,161 patients with type 2diabetes, showed that metformin significantly decreased the risk of developing CRC (relative risk, 0.63; 95% confidence interval,0.50-0.79; P 1⁄4 .001).5 A population-based Taiwanese study of 493,704 men and 502,139 women without CRC at baseline found that metformin users had 27% relative lower risk of developing CRC.

In addition, a recent phase 2 trial study have tested clinically for the very first time, evaluating the efficacy and safety of metformin combined with 5-fluorouracil (5-FU) in patients with progressive and refractory Metastatic colon cancer (Vanessa C, 2016) on the basis of preclinical studies that showed that this combination had synergistic cytotoxicity in CRC and hepatocellular cancer cell lines (Sui x et al, Ling S et al, 2014).

Unfortunately, Despite the indirect evidence that metformin has anti-cancer activity, in several studies, its anti-proliferative effects on cancer patients remain unknown, especially among two populations, the nondiabetic patients, untreated metastatic colon cancer patients (Vanessa C et al, 2016).

Aim of study:

To study the Potential oncological effect augmentation of Metformin addition to standard FOLFOX regimen in non-diabetic metastatic colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

A- •Patients above 18 years old and above B- •Patients who approved to be enrolled in study by documented consent C- Patients with metastatic colon cancer D- NON -Diabetic patients

E- Patients with satisfactory hematological and biochemical functions defined as:

I. Platelets (Plts) >100 x 10^9 II. Creatinine Clearance (Crcl) >60 ml/min or >45-59 but receive single dose of medication III. Aspartate Aminotransferase (AST) AND Alanine Aminotransferases (ALT) <2.5 ULN IV. Absolute Neutrophilic count (ANC) >1,500 / mm^3 V. Eastern Cooperative Oncology Group (ECOG) performance 0-2

Exclusion Criteria:

* Patients with hypersensitivity to metformin, renal or hepatic impairment that may predispose lactic acidosis
* Patients with previous or current severe breathing problems (as obstructive lung disease, severe asthma) or dehydration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate according to Response evaluation criteria in solid tumors ( RECIST) 1.1 | 6 months
  defined as tumor response of patients in Complete remission, partial remission or stable disease from randomization of first subject until database cutoff at 6 month interval
Progression free survival | 1 YEAR

SECONDARY OUTCOMES:
IL-6 Levels | 6 months
  Effect of metformin on IL-6 Levels (from randomization of first subject until database cutoff) at 2 intervals (Baseline - End of study)
Overall Survival | 1 YEAR
  from randomization of first subject until database cutoff / disease progression / death due to any cause) at 2 intervals (Baseline - End of study)
Common terminology criteria adverse events (CTCAE 4.0) | 4 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided